CLINICAL TRIAL: NCT02637206
Title: Skin Irritation Study of GSK2894512 Cream-An Evaluator-Blinded Study to Evaluate the Skin Irritation of GSK2894512 Cream and Placebo Following Single Application by Simple-Patch Test and Photo-Patch Test, and Repeat Application Under Non-occlusive Condition in Healthy Japanese Subjects
Brief Title: Skin Irritation Study of GSK2894512 Cream
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200920
Record Dates: First submitted 2015-09-17; First posted 2015-12-22 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Dermatitis, Atopic
Keywords: Healthy Japanese; GSK2894512; skin safety
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1 (Single Application) (Experimental): All subjects will have two sets (left and right) of 4 semi-occlusive test patches applied to randomized test sites on their upper backs on Day 1. Test patches on left back will be for simple-patch test and those on right back will be for photo-patch test. Each set will consist of approximately 150 micro liter (0.15 mL) of the following study treatments: GSK2894512 0.5% cream, GSK2894512 1% cream, placebo (cream vehicle without the active ingredient) and an empty patch. The test patches will be applied for 24 hrs (photo-patch test) or 48 hrs (simple-patch test).
  Interventions: Drug: GSK2894512 Cream; Drug: Vehicle Cream; Drug: Empty Patch
- Part 2 (Repeat Application) (Experimental): All subjects will have repeat applications of GSK2894512 0.5%, 1% cream and placebo twice a day for 7 days on both side (left and right, 3 in total) of their upper back (approximately 5 centimeter (cm) in diameter >10 cm away from another application area) under non-occlusive conditions and covered with gauze using adhesive. GSK2894512 0.5% and 1% cream and placebo will be randomized according to the randomization code in the same manner as Part 1.
  Interventions: Drug: GSK2894512 Cream; Drug: Vehicle Cream; Drug: Empty Patch

INTERVENTIONS:
Drug: GSK2894512 Cream — GSK2894512 cream supplied will be white to off-white cream packaged in 28-gram laminate tubes of 2 concentrations: 0.5% and 1%, to be applied topically.
Drug: Vehicle Cream — Vehicle Cream (placebo cream without active ingredient) supplied will be white to off-white cream packaged in 28-gram laminate tubes, to be applied topically.
Drug: Empty Patch — Empty patches without any ingredients will be used as negative control.

SUMMARY:
GSK2894512 is a novel anti-inflammatory agent that is currently under development for the topical treatment of atopic dermatitis and chronic plaque psoriasis. This study will be a Phase I, single-center, randomized, partial-blinded (evaluator blinded) study which consists of two parts (Part 1 and 2). Part 1 of this study will assess skin irritation following a single application of GSK2894512 cream at 2 concentrations (e.g. 0.5% and 1%) and placebo by simple-patch test and photo-patch test under semi-occlusive conditions in 20 healthy Japanese volunteers. Part 2 of this study will assess skin irritation following repeat application at 0.5% and 1% of GSK2894512 cream and placebo for 7 days under non-occlusive condition in 6 healthy Japanese volunteers. The study will have Screening visit which will occur within 30 days from the Day 1 visit of each part. Eligible subjects will be able to participate either of Part 1 or Part 2. Subjects will visit the site on Day -1, and hospitalized until the end of all assessments on Day 4 (Part 1) or Day 7 (Part 2). Subjects will re-visit the site on Day 8 (Part 1) or Day 15 (Part 2) for follow-up assessments. This study will be the first to evaluate the safety, tolerability and pharmacokinetics of GSK2894512 cream after single and repeat application in Japanese subjects. Results from this study will enable further clinical investigation in the Japanese population.

ELIGIBILITY:
Inclusion Criteria:

* Japanese males and females aged between 20 and 64 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and 12-lead ECG. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator in consultation with the GlaxoSmithKline (GSK) Medical Monitor if required agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Healthy skin in the potential test site on the back such that erythema and other dermal reactions can be easily visualized.
* Body Mass Index within the range 18.5 - 24.9 kilogram per square meter (kg/m^2,inclusive) and less than 25.0 kg/m^2.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea with simultaneous follicle stimulating hormone (FSH) > 40 milli-international units per milliliter and estradiol < 40 picograms per milliliter (<147 picomole per liter).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form
* Alanine aminotransferase (ALT), alkaline phosphatase and bilirubin <= 1.5x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Based on single QTc values: QT interval corrected for heart rate according to Fridericia's formula (QTcF) < 450 milliseconds; QTcF < 480 msec in subjects with Bundle Branch Block.

Exclusion Criteria:

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of known or suspected intolerance to any of the ingredients of the study products, adhesive tape/plaster, or the test patches.
* Subjects with inherent sensitivity to sun or history of photosensitivity.
* Inability to evaluate the skin at and around the potential test sites on the back due to sunburns, unevenness in skin tone, tattoos, scars, excessive hair, freckles, birthmarks, moles, or other skin damage or abnormality.
* Clinically-relevant skin disease, including psoriasis, eczema, atopic dermatitis, acne, dysplastic nevi, or other skin pathologies, or a history of skin cancer, that may, in the opinion of the investigator, contraindicate participation or interfere with test site evaluations.
* Considered immunocompromised, or has a clinically-relevant history of or currently suffering from any disease or condition that, in the opinion of the investigator, might affect the evaluation of the study product or place the subject at undue risk.
* A positive pre-study syphilis, Hepatitis B surface antigen, Hepatitis C antibody, Human Immunodeficiency Virus antigen antibody or Human T-cell Lymphotropic Virus-1 result of screening.
* A positive pre-study drug screen.
* The subject has donated a unit of blood ">400 milliliter (mL)" within the previous 4 months or ">200 mL" within the previous 1 month prior to the first dosing day.
* The subject has participated in a clinical study with an investigational or a non-investigational drug or device during the previous 4 months prior to the first dosing day.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* The subject planned to concurrently participate in another clinical study or post-marketing study.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 14 days prior to the first application of study medication.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2015-10-27 (Actual); Primary Completion 2015-12-02 (Actual); Study Completion 2015-12-02 (Actual)

PRIMARY OUTCOMES:
Part 1-Positive rate of skin irritability as assessed by simple-patch test following single application of GSK2894512 cream | Up to Day 4
  Each test site for the simple-patch test will be evaluated at 30 minutes (min) and 24 hours (hrs) after removal of medication (48.5 hr and 72 hrs after application, respectively) based on the following criteria proposed by the patch test study group in Japan: no reaction (-); weak erythema (+-); erythema (+); erythema + edema (++); erythema + edema + papules, or vesicles (+++); bullae (++++). Except no reaction (-) and weak erythema (+-), rest all findings from simple-patch test will be considered as positive.
Part 1-Positive rate of photo-urticaria reaction as assessed by photo patch test following single application of GSK2894512 cream | Day 2
  For the photo-patch test, 4 test patches (right back) will be removed 24 hrs after application and the test sites will be exposed to 6.0 joule per square centimeter of ultraviolet A. Each test site will be evaluated at 30 minutes from the irradiation to determine whether there is photo-urticaria or not (i.e positive or negative).
Part 1-Positive rate of photo-toxicity as assessed by photo patch test following single application of GSK2894512 cream | Up to Day 4
  Post photo-urticaria evaluation, the test sites will be re-covered with empty patches, that will be removed at 24 hrs after removal of medication. The test sites will be evaluated at 30 min and 24 hrs after empty patches removal (48.5 and 72 hrs after application, respectively). Assessment Criteria includes: no reaction or similar to the non irradiation site (-); Slightly stronger than the non irradiation site (+-);Definitely stronger than the non irradiation site (+); 2 ranks stronger than the non irradiation site according to the criteria in Japan (++); 3 ranks stronger than the non irradiation site according to the criteria in Japan (+++). Test results of more than or equal to +- will be considered as positive.
Part 2- Positive rate of Skin irritability following repeat application of GSK2894512 cream | Day 1 to Day 8
  Each test site will be evaluated at 30 min after removal of medication based on the following criteria proposed by the patch test study group in Japan: no reaction (-); weak erythema (+-); erythema (+); erythema + edema (++); erythema + edema + papules, or vesicles (+++); bullae (++++). Except no reaction (-) and weak erythema (+-), rest all findings from simple-patch test will be considered as positive.
Part 2- Skin observation (subjective symptom) | Day 1 to Day 7
  At each application site 2 hours following application of study drugs, skin observation (subjective symptom) from application to judgement (2 hours) will be heard from subjects. Symptoms will be recorded as a score ranging from 0-4, where 0=Normal, no discomfort; 1=an awareness, but no discomfort and no intervention required; 2=a noticeable discomfort that causes intermittent awareness; 3=a noticeable discomfort that causes intermittent awareness and interferes occasionally with normal daily activities; 4=a definite continuous discomfort that interferes with normal daily activities.

SECONDARY OUTCOMES:
Part 1: Number of subject with adverse events | From Day 1 to Day 8
  An adverse event (AE) is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Part 2: Number of subject with adverse events | From Day 1 to Day 15
  An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Part 1:Safety as assessed by systolic and diastolic blood pressure measurements | Day -1 to Day 8
  Blood pressure measurements will be measured in supine position after 5 min rest.
Part 2: Safety as assessed by systolic and diastolic blood pressure measurements | Day -1 to Day 15
  Blood pressure measurements will be measured in supine position after 5 min rest.
Part 1:Safety as assessed by pulse rate measurement | Day -1 to Day 8
  Pulse rate measurement will be measured in supine position after 5 min rest.
Part 2: Safety as assessed by pulse rate measurement | Day -1 to Day 15
  Pulse rate measurement will be measured in supine position after 5 min rest.
Part 1:Safety as assessed by12-lead electrocardiogram (ECG) | Day -1 to Day 8
  ECGs will be taken using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and corrected QT and QTc intervals.
Part 2: Safety as assessed by12-lead ECG | Day -1 to Day 15
  ECGs will be taken using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTc intervals.
Part 1:Safety as assessed by clinical laboratory test | Day -1, 4 and 8
  Clinical laboratory parameters include: Hematology, clinical chemistry and urinalysis parameters
Part 2: Safety as assessed by clinical laboratory test | Day -1, 4, 8 and 15
  Clinical laboratory parameters include: Hematology, clinical chemistry and urinalysis parameters
Part 2: Plasma concentration of GSK2894512 | Day 1 and Day 7 (pre-dose, 2, 4 hours post-AM application); Day 3 and Day 5 (pre-dose of AM application)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 200920 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/200920?search=study&search_terms=200920#rs
- Available data/document: Dataset Specification: 200920 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 200920 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 200920 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 200920 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 200920 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 200920 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 200920 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register